CLINICAL TRIAL: NCT02664246
Title: Chinese People's Liberation Army General Hospital
Brief Title: Contrast-induced Nephropathy: Incidence,Risk Factors,Effective Prevention and Management Method
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qian geng, associate chief physician, Chinese PLA General Hospital
Other Study IDs: 16qqy
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Cardio-Renal Syndrome
Keywords: contrast-induced nephropathy; Percutaneous coronary intervention; risk factors; incidence
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: percutaneous coronary intervention

SUMMARY:
This review article have included about ten thousand patients undergoing percutaneous coronary intervention (PCI), aim to identify the incidence of CIN in actual, find some new risk factors and the protecting methods for these factors.

DETAILED DESCRIPTION:
About ten thousand patients undergoing percutaneous coronary intervention (PCI) from 2010 to 2015 are included in this study. We collect the data about the SCr of the patients before and after percutaneous coronary intervention, and define CIN as an increase in SCr of 0.5 mg/dl or 25% from baseline between 48 and 72 h after contrast medium exposure. Besides we obtain the data including clinical characteristics, laboratory data (blood and urine tests) for all the patients. The statistical analysis will find some new risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. congestive heart failure: objective evidences for decreased left ventricular eject fraction (LVEF) <= 50%;
2. moderate to severe chronic kidney disease was defined as an eGFR 15 to 59 mL/min per 1.73 m2, calculated via the abbreviated Modification of Diet in Renal Disease (MDRD) study equation from SCr obtained within 72 hours of enrollment;
3. patients were scheduled to undergo diagnostic cardiac angiography or percutaneous coronary interventions.

Exclusion Criteria:

1. hemodialysis-dependent patients;
2. complicated with severe short-term progressive disease;
3. Patients < 18 years;
4. pregnancy;
5. emergency cardiac catheterisation (eg, primary percutaneous coronary intervention for ST-segment elevation myocardial infarction);
6. exposure to radiographic contrast media within the previous 7 days;
7. acute decompensated heart failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing percutaneous coronary intervention (PCI) from 2010 to 2015
Sampling Method: Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Contrast induced nephropathy postoperation | 7 days
  peak serum creatinine increase of either 0.5 mg/dl or 25% from day 0 through day 7

SECONDARY OUTCOMES:
Composite measure of dialysis or main cardiovascular events | 90 days
  dialysis, myocardial infarction, heart failure and all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Dai Yun Chen, MD, Study Chair — Chinese PLA General Hospital

REFERENCES:
- [Background] Tao SM, Wichmann JL, Schoepf UJ, Fuller SR, Lu GM, Zhang LJ. Contrast-induced nephropathy in CT: incidence, risk factors and strategies for prevention. Eur Radiol. 2016 Sep;26(9):3310-8. doi: 10.1007/s00330-015-4155-8. Epub 2015 Dec 18. PMID 26685852
- [Background] Wichmann JL, Katzberg RW, Litwin SE, Zwerner PL, De Cecco CN, Vogl TJ, Costello P, Schoepf UJ. Contrast-Induced Nephropathy. Circulation. 2015 Nov 17;132(20):1931-6. doi: 10.1161/CIRCULATIONAHA.115.014672. No abstract available. PMID 26572669
- [Background] Andreucci M, Faga T, Pisani A, Sabbatini M, Russo D, Michael A. Prevention of contrast-induced nephropathy through a knowledge of its pathogenesis and risk factors. ScientificWorldJournal. 2014;2014:823169. doi: 10.1155/2014/823169. Epub 2014 Nov 30. PMID 25525625
- [Background] Qian G, Fu Z, Guo J, Cao F, Chen Y. Prevention of Contrast-Induced Nephropathy by Central Venous Pressure-Guided Fluid Administration in Chronic Kidney Disease and Congestive Heart Failure Patients. JACC Cardiovasc Interv. 2016 Jan 11;9(1):89-96. doi: 10.1016/j.jcin.2015.09.026. Epub 2015 Dec 9. PMID 26685074